CLINICAL TRIAL: NCT05208502
Title: Observation of Emergence Time Between Patients Receive General Anesthesia With BIS or 4-channel Spectrogram EEG Monitor
Brief Title: Observational of Emergence Time Between Patients Receive General Anesthesia With BIS or Spectrogram EEG Monitor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201912250RINC
Record Dates: First submitted 2020-06-04; First posted 2022-01-26 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-02

CONDITIONS: General Anesthetic Drug Adverse Reaction; Perioperative/Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BIS: All inclusions will receive the general anesthesia with BIS monitor, a researcher who is not participated in the clinical practice will record the emergence characters and the EEG monitor signal. As the surgery ends, this researcher will record the time started from the end of the surgery to extubation, as well as the emergence quality when the patient was evaluated.
- DSA: All inclusions will receive the general anesthesia with SedLine monitor, a researcher who is not participated in the clinical practice will record the emergence characters and the DSA monitor signal. As the surgery ends, this researcher will record the time started from the end of the surgery to extubation, as well as the emergence quality when the patient was evaluated.
  Interventions: Device: DSA monitor

INTERVENTIONS:
Device: DSA monitor — Next Generation SedLine features an enhanced signal processing engine, which provides processed EEG parameters. This four channel EEG monitor for the monitoring of perioperative anesthesia depth prevent overdose of medication and may help for individualized anesthetic plan
  Other Names: the time when the inclusion started emergence to extubation will be recorded
  Groups: DSA

SUMMARY:
The bispectral index parameter is used to guide the titration of general anesthesia, however; conflicting results between different studies cannot prove the benefit of EEG monitor on improvement of OR efficiency. Next Generation SedLine features an enhanced signal processing engine, which provides processed EEG parameters. This four channel EEG monitor for the monitoring of perioperative anesthesia depth prevent overdose of medication and may help for individualized anesthetic plan. This research intended to observe the emergence time from end of the surgical wound closure to patient awake (or to extubation) with or without SedLine.

DETAILED DESCRIPTION:
This is a clinical observation study. Inclusion criteria are patients with ASA 1-3, age over 20 who need general anesthesia surgery without other neurologic disease. All inclusions will receive the general anesthesia with SedLine monitor, a researcher who is not participated in the clinical practice will record the emergence characters and the EEG monitor signal. The Controls were patients with same criteria without BIS monitor. Sample size was decided if the estimated difference between SedLine group and BIS group are 1 minute and the average estimated as 2 minute. With 80% desired power and default is .05, each group will need 63 cases.

ELIGIBILITY:
Inclusion Criteria:

* patients who need routine general anesthesia
* have no neurological problem
* have no dermo issue over forehead area
* not allergic to the patch

Exclusion Criteria:

* patients who is not agreed

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who need routine general anesthesia
Sampling Method: Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
DSA monitor group has less emergence time | 24 hours
  Patients with SedLine monitor may have shorter emergence time. The prolonged emergence rate is low with SedLine monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Fang Tsai, MD, PhD, Principal Investigator — Operation Theater, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan